CLINICAL TRIAL: NCT04658472
Title: A Phase 2, Multicenter, Open-label, Non-randomized, Proof-of-concept Study Evaluating the Efficacy, Safety, and Tolerability of SAR445088 in Adults With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: Proof-of-concept Study for SAR445088 in Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDY16744; U1111-1246-7023 (Registry Identifier: ICTRP); 2024-512345-16 (Registry Identifier: CTIS); 2020-004006-54 (EudraCT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SOC-Refractory Initial Dose (Experimental): Part A: Eligible participants will receive SAR445088 for 24 weeks. Participants who do not enroll into Part B will be asked to attend a final safety follow-up visit that will take place 22 weeks after Week 24 (approximately (~)at Week 46).
  Part B: Participants who successfully complete Part A, will be reassessed for continuing eligibility and will be given the option of rolling into Part B, where they will continue receiving SAR445088 for an additional 52 weeks. At the end of the Part B treatment period, participants will be asked to attend a safety follow-up visit that will take place 22 weeks after the last SAR445088 dose (approximately week 98) if they will not continue in Part C.
  Part C: Participants from Part B who enter Part C will continue receiving SAR445088 until the end of study.
  Participants who discontinue at any time during Part C will be asked to attend a safety follow-up visit that will take place 22 weeks after the last SAR445088 dose.
  Interventions: Drug: SAR445088 (IV); Drug: SAR445088 (SC)
- SOC-Refractory Low Dose (Experimental): Part A: Eligible participants will receive SAR445088 for 24 weeks. Participants who do not enroll into Part B will be asked to attend a final safety follow-up visit that will take place 22 weeks after Week 24 (approximately at Week 46).
  Part B: Participants who successfully complete Part A, will be reassessed for continued eligibility and will be given the option to roll into Part B, where they will continue receiving SAR445088 for an additional 52 weeks. At the end of the Part B treatment period, participants will be asked to attend a safety follow-up visit that will take place 22 weeks after the last SAR445088 dose (approximately week 98) if they do not continue in Part C.
  Part C: Participants from Part B who enter Part C will continue receiving SAR445088 until the end of study.
  Participants who discontinue at any time during Part C will be asked to attend a safety follow-up visit that will take place 22 weeks after the last SAR445088 dose.
  Interventions: Drug: SAR445088 (IV); Drug: SAR445088 (SC)
- SOC-Treated Initial Dose (Experimental): Part A: Eligible participants will receive SAR445088 for 24 weeks. Weeks 1-12 (overlap period): Participants will be given SAR445088 with superimposing effects of SOC therapy; Weeks 13-24: SAR445088 given.
  Participants who do not enroll into Part B will attend final safety follow-up visit at 22 weeks after Week 24 (~Week 46).
  Part B: Participants who successfully complete Part A, will be reassessed for continuing eligibility and will be given option of rolling into Part B, and continue receiving SAR445088 for 52 weeks. At the end of the Part B treatment period, participants will be asked to attend a safety follow-up visit that will take place 22 weeks after the last SAR445088 dose (~week 98) if they do not continue in Part C.
  Part C: Participants from Part B who enter Part C will continue receiving SAR445088 until end of study.
  Participants who discontinue at any time during Part C will be asked to attend a safety follow-up visit at 22 weeks after the last SAR445088 dose.
  Interventions: Drug: SAR445088 (IV); Drug: SAR445088 (SC)
- SOC-Naive (Experimental): Part A: Eligible participants will receive SAR445088 for 24 weeks. Participants who do not enroll into Part B will be asked to attend a final safety follow-up visit that will take place 22 weeks after Week 24 (approximately at Week 46).
  Part B: Participants who successfully complete Part A, will be reassessed for continuing eligibility and will be given the option of rolling into Part B, where they will continue receiving SAR445088 for an additional 52 weeks. At the end of the Part B treatment period, participants will be asked to attend a safety follow-up visit that will take place 22 weeks after last SAR445088 dose (approximately week 98) if they do not continue in Part C.
  Part C: Participants from Part B who enter Part C will continue receiving SAR445088 until the end of study. Participants who discontinue at any time during Part C will be asked to attend a safety follow-up visit that will take place 22 weeks after last SAR445088 dose.
  Interventions: Drug: SAR445088 (IV); Drug: SAR445088 (SC)
- SOC-Treated Low Dose (Experimental): Part A: Eligible participants will receive SAR445088 for 24 weeks. Weeks 1-12 (overlap period): Participants will be given SAR445088 with superimposing effects SOC therapy; Weeks 13-24: SAR445088. Participants who do not enroll into Part B will attend a final safety follow-up visit that will take place 22 weeks after Week 24 (~Week 46).
  Part B: Participants who successfully complete Part A, will be reassessed for continued eligibility, will be given the option of rolling into Part B, and continue receiving SAR445088 for 52 weeks. At the end of the Part B treatment period, participants will attend a safety follow-up visit that will take place 22 weeks after the last SAR445088 dose (~week 98) if they do not continue in Part C.
  Part C: Participants from Part B who enter Part C will continue receiving SAR445088 until end of study. Participants who discontinue at any time in Part C will attend a safety follow-up visit that will take place 22 weeks after the last SAR445088 dose.
  Interventions: Drug: SAR445088 (IV); Drug: SAR445088 (SC)

INTERVENTIONS:
Drug: SAR445088 (IV) — Pharmaceutical form: Solution for Injection Route of Administration: Intravenous (IV)
Drug: SAR445088 (SC) — Pharmaceutical form: Solution for Injection Route of Administration: Subcutaneous (SC)

SUMMARY:
Primary Objectives:

* Part A: Efficacy of SAR445088 across three subpopulations of CIDP patients: standard of care (SOC)-Treated, SOC-Refractory and SOC-Naive
* Part B:Long-term safety and tolerability of SAR445088 in CIDP

Secondary Objectives:

* Part A:

  * Safety and tolerability of SAR445088 in CIDP
  * Immunogenicity of SAR445088
  * Efficacy of SAR445088 with overlapping SOC (SOC-Treated group)
* Part B:

  * Durability of efficacy during long-term treatment with SAR445088 in CIDP
  * Long-term immunogenicity of SAR445088 in CIDP

DETAILED DESCRIPTION:
The duration of the study for a participant will include:

Part A Screening period: up to 6 weeks. Treatment period: once successfully screened, enrolled participants will receive study intervention for 24 weeks.

Safety follow-up visit: participants who do not enroll (rollover) into Part B will be asked to attend a final safety follow-up visit that will take place 22 weeks after Week 24, ie, approximately at Week 46.

Part B Treatment period (extension): for all groups, this period will consist of 52 weeks of treatment with SAR445088 (Weeks 24 to 76; Part A and B total treatment period of 76 weeks).

Safety follow-up visit: participants who do not enroll (rollover) into Part C will be asked to attend a safety follow-up visit that will take place 22 weeks after the last SAR445088 dose (Week 98).

Part C Treatment period: participants who complete Part B will be reassessed for continuing eligibility, defined as having successfully completed Part B (received IMP until the Week 76 visit and have responded to SAR445088 based on Investigator's medical judgement), with no new safety concerns. Eligible participants will be given the option of rolling into Part C, where they will continue receiving SAR445088 until end of study.

End of study has been defined as the last safety follow-up visit for the last patient which occurs 22 weeks after last dose.

In addition, there is a follow-up call 56 weeks ±14 days after last dose to confirm negative result of urine pregnancy test for women of childbearing potential who are participating in the study, or to query male participants regarding pregnancy of partners who are women of childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age at the time of signing the informed consent.
* Documented definite or probable diagnosis of CIDP (typical CIDP, pure motor CIDP, or Lewis-Sumner Syndrome) according to the European Federation of Neurological Societies (EFNS)/Peripheral Nerve Society (PNS) Task Force first revision.
* Belonging to one of the following three groups: standard-of-care (SOC)-Treated, SOC-Refractory or SOC-Naive, as defined below.
* SOC-Treated (all criteria a-c must be met): a) Documented evidence of objective response to SOC, with clinically meaningful improvement. Clinically meaningful improvement is defined as one of the following: ≥1-point decrease in adjusted INCAT score, ≥4 points increase in RODS total score, ≥3 points increase in MRC Sum score, ≥8 kilopascal improvement in mean grip strength (one hand), or an equivalent improvement based on information documented in medical records and per the PI's judgement. b) Must be on stable SOC therapy, defined as no change greater than 10% in frequency or dose of immunoglobulin therapy or corticosteroids within 8 weeks prior to screening, remaining at stable SOC therapy until the time of first SAR445088 dosing. c) Evidence of clinically meaningful deterioration on interruption or dose reduction of SOC therapy within 24 months prior to screening, determined by clinical examination or medical records. Clinically meaningful deterioration is defined as one of the following: ≥1-point increase in adjusted INCAT score, decrease in RODS total score ≥4 points, decrease in MRC Sum score ≥3, mean grip strength worsening of ≥8 kilopascals (one hand), or an equivalent deterioration based on information from medical records and at the PI's judgement.
* SOC-Refractory (all criteria a-d must be met): a) Evidence of failure or inadequate response to SOC defined as no clinically meaningful improvement and persistent INCAT score ≥2 after treatment for a minimum of 12 weeks on SOC prior to screening. A clinically meaningful improvement is defined as one of the following: ≥1-point decrease in adjusted INCAT score, increase in RODS total score ≥4 points, increase in MRC Sum score ≥3, mean grip strength improvement of ≥8 kilopascals (one hand), or equivalent improvement based on information from medical records and at the PI's judgement.

Or

* Unable to receive or continue treatment with immunoglobulins or corticosteroids due to side effects.
* b) Patient has not received immunoglobulins (IVIg or SCIg) within 12 weeks prior to screening. c) Certain immunosuppressant drugs are allowed in this group if taken for ≥6 months and at a stable dose for ≥3 months prior to screening: azathioprine, methotrexate, mycophenolate mofetil and cyclosporine. Oral corticosteroids are allowed if on a stable dose of <20 mg/day of prednisone (or equivalent dose for other oral corticosteroids) for ≥3 months prior to screening. d) INCAT score: 2-9 (a score of 2 should be exclusively from leg disability component of INCAT).
* SOC-Naive (all criteria a-c must be met): a) Participants without previous treatment for CIDP or participants who received immunoglobulins (IVIg or SCIg) or corticosteroids but were stopped for reasons other than lack of response or side effects. b) Not treated with immunoglobulins (IVIg or SCIg) or corticosteroids for at least 6 months prior to screening. c) INCAT score: 2-9 (a score of 2 should be exclusively from leg disability component of INCAT.
* Documented vaccinations against encapsulated bacterial pathogens given within 5 years of enrollment or initiated a minimum of 14 days prior to first dose
* A female participant must use a double contraception method including a highly effective method of birth control from inclusion and up to 52 weeks plus 30 days after the last study dose and agree not to donate eggs, ova or oocytes during this period.
* A female participant must have a negative highly sensitive pregnancy test (urine or serum) as required by local regulations within 24 hours before the first dose of study intervention.
* Male participants, whose partners are of childbearing potential must accept to use, during sexual intercourse, a double contraceptive method according to the following: condom plus an additional highly effective contraception
* Male participants must have agreed not to donate sperm during the intervention and up to 52 weeks after the last dose.
* Capable of giving signed informed consent

Exclusion Criteria:

* Polyneuropathy of other causes, including but not limited to hereditary demyelinating neuropathies, neuropathies secondary to infection or systemic disease, diabetic neuropathy, drug- or toxin-induced neuropathies, multifocal motor neuropathy, polyneuropathy related to IgM monoclonal gammopathy, POEMS syndrome, lumbosacral radiculoplexus neuropathy, pure sensory CIDP and acquired demyelinating symmetric (DADS) neuropathy (also known as distal CIDP).
* Any other neurological or systemic disease that can cause symptoms and signs interfering with treatment or outcome assessments.
* Poorly controlled diabetes (HbA1c >7%).
* Serious infections requiring hospitalization within 30 days prior to screening and any active infection requiring treatment during screening.
* Clinical diagnosis of SLE.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study. Specifically, history of any hypersensitivity reaction to SAR445088 or its components or of a severe allergic or anaphylactic reaction to any humanized or murine monoclonal antibody.
* Participants with a history of suicidality in the six months prior to screening or currently at risk of committing suicide.
* Presence of conditions (medical history or laboratory assessments) that may predispose the participant to excessive bleeding or increased risk of infection.
* Evidence of CIDP relapse within 6 weeks after receiving a vaccination.
* Recent or planned major surgery that could confound the results of the trial or put the participant at undue risk.
* Treatment with plasma exchange within 12 weeks prior to screening.
* Prior treatment with rituximab or ocrelizumab in the 6 months prior to SAR445088 dosing or until return of B-cell counts to normal levels, whichever is longer.
* Immunosuppressive/chemotherapeutic medications such as azathioprine, methotrexate, cyclophosphamide, cyclosporine, mycophenolate mofetil, tacrolimus, interferon, TNF-alpha inhibitor: within 6 months prior to dosing (except for some cases as indicated in the SOC-Refractory group).
* Treatment (any time) with highly immunosuppressive/chemotherapeutic medications with sustained effects, eg, mitoxantrone, alemtuzumab, cladribine.
* Treatment (any time) with total lymphoid irradiation or bone marrow transplantation.
* Use of any specific complement system inhibitor (eg, eculizumab) within 12 weeks or 5 times the half-life of the product, whichever is longer, prior to screening.
* Pregnant (defined as positive β-HCG blood test) or lactating females.
* Positive result on any of the following tests: hepatitis B surface (HBsAg) antigen, anti-hepatitis B core antibodies (anti-HBc Ab)-unless anti-hepatitis B surface antibodies (anti-HBs Ab) are also positive , indicating natural immunity-, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 antibodies).
* Evidence of IgG4 autoantibodies against paranodal proteins (NF155 and CNTN1).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Part A, SOC-Treated: Percentage of participants relapsing after withdrawal of SOC and during the SAR445088 treatment period | Day 1 up to 24 weeks
  Relapse will be defined as ≥1-point increase in adjusted Inflammatory neuropathy cause and treatment (INCAT) disability score. The Investigator/rater will evaluate the level of impairment in participants? arms and legs each on a scale of 0 (least impaired) to 5 (most impaired), in the context of a neurological examination, and will record the added scores (range 0 to 10) per the INCAT reporting instructions. A low score reflects no or minimal disability eg, no arm dysfunction or walking normally, whereas higher scores indicate more disability eg, wheelchair bound or no purposeful arm movement.
Part A, SOC-Refractory (initial and low dose group) and SOC-Naive: Percentage of participants responding during the SAR445088 treatment period | Day 1 up to 24 weeks
  Response will be defined as ≥1-point decrease in adjusted INCAT disability score. The Investigator/rater will evaluate the level of impairment in participants? arms and legs each on a scale of 0 (least impaired) to 5 (most impaired), in the context of a neurological examination, and will record the added scores (range 0 to 10) per the INCAT reporting instructions. A low score reflects no or minimal disability eg, no arm dysfunction or walking normally, whereas higher scores indicate more disability eg, wheelchair bound or no purposeful arm movement.
Part B: Number of participants reported with adverse events | Day 1 up to Week 98
  Number of participants reported with adverse events during 76 weeks of treatment and 22 weeks of follow-up.

SECONDARY OUTCOMES:
Part A: Number of participants reported with adverse events | Day 1 up to 46 Weeks
  Number of participants reported with adverse events during 24 weeks of treatment period and if not enrolled to Part B, 22 weeks of follow-up period.
Part A: Number of participants with incidence and titer of anti-SAR445088 antibodies (ADA) | Day 1 up to 46 Weeks
  Incidence and titer of anti-SAR445088 antibodies (ADA) will be assessed during the 24 weeks of treatment period and if not enrolled to Part B, 22 weeks of follow-up period.
Part A: Percentage of participants in the SOC-Treated group improving during the overlap treatment period | Day 1 up to 12 Weeks
  Improvement will be defined as ≥1 point decrease in adjusted INCAT disability score. The Investigator/rater will evaluate the level of impairment in participants? arms and legs each on a scale of 0 (least impaired) to 5 (most impaired), in the context of a neurological examination, and will record the added scores (range 0 to 10) per the INCAT reporting instructions. A low score reflects no or minimal disability eg, no arm dysfunction or walking normally, whereas higher scores indicate more disability eg, wheelchair bound or no purposeful arm movement.
Part B, SOC-Treated (initial dose group): Percentage of participants relapse-free during the treatment extension period | Week 24 up to Week 76
  Relapse-free will be defined as no increase in adjusted INCAT disability score >2 points. The Investigator/rater will evaluate the level of impairment in participants? arms and legs each on a scale of 0 (least impaired) to 5 (most impaired), in the context of a neurological examination, and will record the added scores (range 0 to 10) per the INCAT reporting instructions. A low score reflects no or minimal disability eg, no arm dysfunction or walking normally, whereas higher scores indicate more disability eg, wheelchair bound or no purposeful arm movement.
Part B, SOC-Refractory (initial and low dose group) and SOC-Naive: Percentage of participants with sustained response during the treatment extension period | Week 24 up to Week 76
  Maintenance of response will be defined as no increase in adjusted INCAT disability score greater than or equal to 2 points. The Investigator/rater will evaluate the level of impairment in participants arms and legs each on a scale of 0 (least impaired) to 5 (most impaired), in the context of a neurological examination, and will record the added scores (range 0 to 10) per the INCAT reporting instructions. A low score reflects no or minimal disability eg, no arm dysfunction or walking normally, whereas higher scores indicate more disability eg, wheelchair bound or no purposeful arm movement.
Part B: Long-term immunogenicity | Day 1 Up to Week 98
  Incidence and titer of anti-SAR445088 antibodies during the entire SAR445088 treatment period and follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (32):
- United States (5):
  - University of Southern California Site Number : 8400004, Los Angeles, California
  - University of California Irvine Site Number : 8400002, Orange, California
  - The University of Kansas Clinical Research Center Site Number : 8400003, Fairway, Kansas
  - University of Minnesota Site Number : 8400006, Minneapolis, Minnesota
  - Columbia University Site Number : 8400005, New York, New York
- Canada (2):
  - Investigational Site Number : 1240001, Gatineau, Quebec
  - Investigational Site Number : 1240002, Québec
- China (3):
  - Investigational Site Number : 1560002, Fuzhou
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560004, Wuhan
- France (5):
  - Investigational Site Number : 2500003, Bordeaux
  - Investigational Site Number : 2500004, Garches
  - Investigational Site Number : 2500005, Le Kremlin-Bicêtre
  - Investigational Site Number : 2500001, Marseille
  - Investigational Site Number : 2500002, Nice
- Germany (4):
  - Investigational Site Number : 2760001, Düsseldorf
  - Investigational Site Number : 2760003, Essen
  - Investigational Site Number : 2760002, Göttingen
  - Investigational Site Number : 2760004, Tübingen
- Italy (4):
  - Investigational Site Number : 3800002, Rome, Lazio
  - Investigational Site Number : 3800005, Rozzano, Milano
  - Investigational Site Number : 3800003, Genova
  - Investigational Site Number : 3800001, Milan
- Netherlands (2):
  - Investigational Site Number : 5280001, Amsterdam
  - Investigational Site Number : 5280002, Utrecht
- Investigational Site Number : 6160001, Lublin, Lublin Voivodeship, Poland
- Serbia (3):
  - Investigational Site Number : 6880001, Belgrade
  - Investigational Site Number : 6880002, Belgrade
  - Investigational Site Number : 6880003, Niš
- Spain (3):
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Querol L, Lewis RA, Hartung HP, Van Doorn PA, Wallstroem E, Luo X, Alonso-Alonso M, Atassi N, Hughes RAC. An innovative phase 2 proof-of-concept trial design to evaluate SAR445088, a monoclonal antibody targeting complement C1s in chronic inflammatory demyelinating polyneuropathy. J Peripher Nerv Syst. 2023 Jun;28(2):276-285. doi: 10.1111/jns.12551. Epub 2023 May 31. PMID 37119056
- See also: PDY16744 Plain Language Results Summaries — https://www.trialsummaries.com/Study/StudyDetails?id=25317&tenant=MT_SNY_9011